CLINICAL TRIAL: NCT02298075
Title: Response Rate and Response Duration After Discontinuation of Treatment With Thrombopoietin Receptor Agonists in Patients Affected by Primary Immune Thrombocytopenia (pITP): Retrospective Study
Brief Title: Response Rate and Duration After Discontinuation Thrombopoietin Receptor Agonists Primary Immune Thrombocytopenia
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: ITP0714
Record Dates: First submitted 2014-11-17; First posted 2014-11-21 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Immune Thrombocytopenia
Keywords: Immune thrombocytopenia; Primary; Thrombopoietin receptor agonist
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Eltrombopag — Investigation of the impact of TPO-RAs on the achievement of sustained and persistent response after discontinuation in adult patients affected by pITP.
  Other Names: Thrombopoietin Receptor Agonists (TPO-RAs)
Drug: Romiplostin — Investigation of the impact of TPO-RAs on the achievement of sustained and persistent response after discontinuation in adult patients affected by pITP.
  Other Names: Thrombopoietin Receptor Agonists (TPO-RAs)

SUMMARY:
The primary objective of the study is the evaluation of sustained response rate after discontinuation of treatment with TPO-RAs, Eltrombopag and Romiplostim, in persistent or chronic pITP patients who failed one or more therapy lines, splenectomy included.

DETAILED DESCRIPTION:
Increasing evidence exists in the literature on the persistent response after TPO-RAs discontinuation. However, the available data consist of description of case reports from different patients' series. At this time, systematic data collections on this topic do not exist and the real incidence of such persistent response is unknown. Therefore, because of the increasing interest in this new and challenging therapeutic field, also for the therapeutic implications, we would like to investigate the impact of TPO- RAs on the achievement of sustained and persistent responses after their discontinuation in the Italian adult patients affected by pITP who have been referred to the GIMEMA Centers.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent according to ICH/EU/GCP and national local laws;
* Persistent or chronic pITP adult patients who have been treated with TPO-RAs therapy after failure of one or more therapy lines, splenectomy included;
* Age > 18 years.

Exclusion Criteria:

* Active malignancy;
* Active malignancy;
* HCVAb, HIVAb, HBsAg, HBcAb seropositive status;
* Chronic liver disease;
* Treatment with Rituximab less than 8 weeks before TPO-RAs start;
* Recent splenectomy (less than 8 weeks) before TPO-RAs start. Active malignancy;
* HCVAb, HIVAb, HBsAg, HBcAb seropositive status;
* Chronic liver disease;
* Treatment with Rituximab less than 8 weeks before TPO-RAs start;
* Recent splenectomy (less than 8 weeks) before TPO-RAs start. HCVAb, HIVAb, HBsAg, HBcAb seropositive status;
* Chronic liver disease;
* Treatment with Rituximab less than 8 weeks before TPO-RAs start;
* Recent splenectomy (less than 8 weeks) before TPO-RAs start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by primary immune thrombocytopenia (pITP)
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2016-04; Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Estimation of sustained response rate after discontinuation of treatment with TPO-RAs in terms of patients still alive in Complete Response or R at more than 4 weeks after discontinuation. | One year from start of recruitment.

SECONDARY OUTCOMES:
Frequency of the type of response in patients treated with TPO-RAs in absence of concomitant or rescue medication, in order to estimate the rate of Response (R) and Complete Response (CR). | One year from start of recruitment.
Estimation of the suspension criteria in terms of frequency of discontinuation causes for each center. | One year from start of recruitment.
Estimation of the duration of sustained response in terms of patients alive in CR or R at 6 and 12 months after sustained response achievement. | One year from start of recruitment.
Estimation of incidence of relapse and loss of response at 6 and 12 months after sustained response achievement. | One year from start of recruitment.
Estimation of treatment duration starting from the date of first dose of TPO-RAs. | One year from start of recruitment.
Description of Platelet levels and TPO-RAs dosage at stop. | One year from start of recruitment.
Description of patients' characteristics in term of: biological and clinical features, disease duration at the beginning of TPO-RAs, number and type of therapy lines preceding TPO-RAs treatment, platelet levels at TPO-RAs start. | One year from start of recruitment.
Assessment of an association between previous splenectomy and sustained response after discontinuation of treatment with TPO-RAs. | One year from start of recruitment.
Description of concomitant therapies since TPO-RAs start in terms of type and duration of therapies. | One year from start of recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gabriella Mazzucconi, Study Chair — Policlinico Umberto I, Hematology Department.
Locations (13):
- Italy (13):
  - S.O.C. di Medicina Interna B - Ospedale - Cardinal Massaia di Asti, Asti
  - Istituto di Ematologia "Lorenzo e A. Seragnoli", Bologna
  - Unità di Onco-Ematologia - Azienda Ospedaliera - Garibaldi, Catania
  - Unità di Ricerca e di Malattie del sangue - Ematologia San Luca Vecchio Pad. 16 - 1° Piano, Florence
  - Clinica Medica III - Padiglione ex isolamento - Azienda Ospedale Università San Martino, Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Azienda Ospedaliera "S.Gerardo", Monza
  - Ematologia - Ospedale San Carlo, Potenza
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - U.O.C. Ematologia - Ospedale S. Eugenio, Rome
  - Università degli studi "Sapienza" di Roma, Rome
  - Ematologia - Dipartimento di Medicina Clinica e Sperimentale, Sassari

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it